CLINICAL TRIAL: NCT06919003
Title: Improving Deceased-Donor Kidney Transplant Outcomes Via a Single Intragraft Injection of C1 Esterase Inhibitor (RTB-021)
Brief Title: Improving Deceased-Donor Kidney Transplant Outcomes Via a Single Intragraft Injection of C1 Esterase Inhibitor (IMPROVE TRIAL)
Acronym: IMPROVE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT RTB-021
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Kidney Transplant
Keywords: Kidney transplant; Deceased donor; Intragraft injection; C1 esterase inhibitor
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — Complement C1 Inhibitor Protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This study is a double-blind, placebo-controlled study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Berinert (Experimental)
  Interventions: Biological: Berinert
- Saline (Placebo Comparator)
  Interventions: Other: Placebo for Berinert

INTERVENTIONS:
Biological: Berinert — Administered as a 10 ml renal artery infusion approximately 1-2 hours before implantation and reperfusion of the allograft
  Other Names: C1 esterase inhibitor; C1INH
  Arms: Berinert
Other: Placebo for Berinert — Administered as a 10 ml renal artery infusion approximately 1-2 hours before implantation and reperfusion of the allograft
  Arms: Saline

SUMMARY:
The purpose of this study is to find out if Berinert can improve kidney function in the first year after transplant and to find out what effects, good or bad, Berinert will have in the kidney recipient. This research study will compare Berinert to placebo. The placebo looks exactly like Berinert but does not contain any active drug. Placebos are used in research studies to see if the results are due to the study drug or due to other reasons. Neither you or the study doctor can choose or know which group is assigned.

The primary objective is to test whether intrarenal artery C1 esterase inhibitor (C1INH) injection into the donor kidney prior to transplantation improves kidney function in recipients of high risk, deceased donor kidney transplants as measured by 12-month Estimated Glomerular Filtration Rate (eGFR) Chronic Kidney Disease Epidemiology Collaboration (CDK-EPI)

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be able to understand and provide informed consent
2. Adults who are on chronic dialysis therapy and are on the wait list for deceased donor kidney transplant
3. Recipients who are ABO compatible with donor allograft
4. Negative crossmatch and no donor specific anti-HLA antibody (DSA) on most recent pretransplant serum sample as determined by local site
5. Female participants of childbearing potential must have a negative pregnancy test upon study entry
6. All participants with reproductive potential must agree to use highly effective contraception for at least 12-moths post-transplant. Oral estrogen containing contraception must not be used during the first 3 months post-transplant
7. Hepatitis C Virus Ab positive participants with negative Hepatitis C virus (HCV) Polymerase chain reaction (PCR) are eligible if they have spontaneously cleared infection or are in sustained virologic remission
8. Hepatitis C Virus negative recipients of a Hepatitis C Virus positive organ are eligible if they will be treated with the intent of inducing a sustained virologic remission
9. Recipients of kidneys arriving to the transplant center on ex vivo hypothermic machine perfusion pumps are eligible
10. Vaccines up to date per Division of Allergy, Immunology, and Transplantation (DAIT) guidance for patients in transplant trials
11. Anticipated Cold Ischemia Time (CIT) >=12 hours
12. Kidney Donor Profile Index (KDPI) 21-95%. For KDPI 21-34% to be eligible, anticipated CIT must be >=24 hours
13. Patients with normal coagulation

Exclusion Criteria:

1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol
2. Any prior or concurrent non-renal solid organ, or cellular transplant, or waitlisted for multi-organ transplant
3. Patients receiving enbloc kidneys
4. Kidneys receiving normothermic perfusion
5. Patients with a known pro-thrombotic disorder
6. Patients with a history of thrombosis or hyper-coagulable state, excluding dialysis access clotting
7. Body mass index (BMI) >=40 kg/m^2
8. Patients with a history of Hereditary Angioedema or use of C1 esterase inhibitor (C1INH) containing products or recombinant C1INH within 15 days prior to study entry
9. Patients with a known hypersensitivity to treatment with Berinert
10. Patients requiring chronic anti-coagulation or anti-platelet therapy. ASA and NSAIDS are allowed
11. Presence of active malignancy or history of malignancy less than 5 years in remission, excluding adequately treated in-situ cervical carcinoma, low grade prostate carcinoma, or adequately treated basal or squamous cell carcinoma of the skin
12. Patients who are positive for Hep B infection (Hepatitis B surface antigen (HBsAg)+ or anti-HBcore +)
13. Any active infection
14. Human immunodeficiency virus (HIV) infection
15. Enrollment in another investigational trial
16. Recent recipient of any licensed or investigational live attenuated vaccine(s) within 4 weeks of enrollment
17. Current or planned use of immunomodulatory agents including but not limited to rituximab, belatacept, eculizumab, JAK inhibitors, anti-TNF agents
18. Female participants who are pregnant or lactating
19. Past or current medical problems, inclusive of mental health and substance abuse concerns, or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2031-05-30 (Estimated); Study Completion 2032-05-30 (Estimated)

PRIMARY OUTCOMES:
Difference between study arms in renal function | At 12-months post-transplantation
  Measured as Estimated Glomerular Filtration Rate Chronic Kidney Disease Epidemiology Collaboration (eGFRCKD-EPI) in ml/min/1.73m^2

SECONDARY OUTCOMES:
Comparison between the treated and control group of the full iBox score | At 12-months post-transplantation
  The iBox scoring system is a composite biomarker panel. The full iBox scoring system consists of 4 elements all obtained 1-year post-transplant: a) eGFR (MDRD), b) DSA, c) urinary protein/creatine ratio, and d) histological abnormalities on a surveillance biopsy.
Incidence of biopsy proven acute rejection (BPAR) | At 12-months post-transplantation
Incidence of proteinuria | At 12-months post-transplantation
  Measured as spot urine protein/creatinine >1 g/g
Incidence of de novo donor specific anti-Human Leukocyte Antigen (HLA) antibody (DSA) | At 12-months post-transplantation
  Defined as the incidence of de novo DSA on standard of care or protocol directed blood draws up to and including the 12-month protocol blood draw.
Incidence of Grade 3 or higher infections | At 12-months post-transplantation
Incidence of Grade 3 or higher intraoperative or postoperative hemorrhage | Within 4 weeks after transplantation
Incidence of thrombotic or thromboembolic events | Within 4 weeks after transplantation
  Excluding superficial thrombophlebitis, catheter-related thrombosis and dialysis access thrombosis
Incidence of T cell mediated rejection (TCMR) that is steroid resistant | At 12-months post-transplantation
Incidence of TCMR that is BANFF grade 2 or higher | At 12-months post-transplantation
Incidence of antibody mediated rejection (ABMR) | At 12-months post-transplantation
Incidence of death | At 12-months post-transplantation
Incidence of Graft loss (including primary non function) | At 12-months post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Heeger, MD, Study Chair — Cedars-Sinai Medical Center; Sindhu Chandran, MBBS, MD, Study Chair — Cedars-Sinai Medical Center; Stanley Jordan, MD, Study Chair — Cedars-Sinai Medical Center
Locations (4):
- United States (4):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — http://www.niaid.nih.gov/about/dait